CLINICAL TRIAL: NCT04397107
Title: The Therapeutic Value and Mechanism of Recombinant Human Interleukin-2 on Children With Rheumatic Diseases (Systemic Lupus Erythematosus, Primary Sjögren Syndrome, Juvenile Idiopathic Arthritis)
Brief Title: The Therapeutic Value and Mechanism of Recombinant Human Interleukin-2 on Children With Rheumatic Diseases
Acronym: SLE，pSS，JIA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The First Hospital of Jilin University (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 20K013-001
Record Dates: First submitted 2020-05-06; First posted 2020-05-21 (Actual); Last update posted 2022-08-18 (Actual); Status verified 2022-08

CONDITIONS: Systemic Lupus Erythematosus
MeSH Terms: conditions — Lupus Erythematosus, Systemic | interventions — Interleukin-2; aldesleukin; Injections

STUDY DESIGN:
Intervention Model Description: One group patients were treated with IL-2 and another group patients were treated with routine therapy.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Recombinant Human Interleukin-2 (Experimental): Induced remission period,recombinant human IL-2(500,000 unit per square meter) infusions five days;Maintenance treatment period,recombinant human IL-2 infusions five days then once every two weeks for 6 months.
  Interventions: Drug: IL-2
- Traditional therapy (No Intervention): Patients were treated with glucocorticoid and/or immunosuppressor.

INTERVENTIONS:
Drug: IL-2 — Patients were received low dose recombinant human Interleukin-2
  Other Names: Recombinant Human Interleukin-2 for Injection
  Arms: Recombinant Human Interleukin-2

SUMMARY:
The study aims to explore the therapeutic value and mechanism of Interleukin-2 on children with rheumatic diseases (Systemic Lupus Erythematosus, Primary Sjögren Syndrome, Juvenile Idiopathic Arthritis).

DETAILED DESCRIPTION:
The investigators designed a single center, open-label, prospective study that routinely administered low-dose IL-2 therapy to monitor the improvement of clinical and laboratory parameters to explore its efficacy and to observe changes in immune cell subsets and cytokines.

Methods: Patients were divided into two groups. One received standard therapy, while another one administrate with low-does IL-2 plus standard therapy.

ELIGIBILITY:
Inclusion Criteria:

1. age <18 years old
2. meet the diagnostic criteria of disease classification
3. HIV negative;Negative for Hepatitis B Virus and Hepatitis C Virus.

Exclusion Criteria:

1. heart failure (cardiac function ≥ grade III NYHA)
2. liver insufficiency (upper limit of normal range of transaminase > 2 times)
3. renal insufficiency (creatinine clearance ≤30ml/min)
4. acute or severe infections such as bacteremia and sepsis
5. malignant tumor
6. high-dose steroid pulse therapy or intravenous injection of glucocorticoids in the last 1 month;Rituximab, infliximab or other biological agents were used
7. mental disorders or any other chronic illness or substance abuse may interfere with the ability to comply with agreements or provide information
8. Inability to comply with IL-2 treatment regimen.

Max Age: 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 46 (Actual)
Dates: Start 2020-08-15 (Actual); Primary Completion 2022-05-31 (Actual); Study Completion 2022-06-30 (Actual)

PRIMARY OUTCOMES:
Change in steroid dose and immunosuppressor dose at 1 year compared to control group | 1 year
  The average daily doses of steroid and immunosuppressor per square meter was recorded

SECONDARY OUTCOMES:
The Immunologic Impact of IL-2 Treatment | 1 month,3 month,6 month,1 year
  Laboratory measures were detected, including, C3, C4 and anti-dsDNA titres.
Immunological Responses | 1 month,3 month,6 month,1 year
  Enumeration of the number of subjects with a change in the absolute number of immune cells and serum cytokines in the peripheral blood
Change from baseline in SELENA SLEDAI Score | 1 month,3 month,6 month,1 year
  Assessment version of the SLE Disease Activity Index (SELENA-SLEDAI) change. The higher the score represent the worse of the disease. The total score ranges from 0 to 105 points.
Change from baseline in EULAR SS disease activity index | 1 month,3 month,6 month,1 year
  Low-activity (ESSDAI<5),moderate-activity (5≤ESSDAI≤13) ,high-activity (ESSDAI≥14) levels.
Incidence of adverse drug reactions | up to 1 year
  Adverse events includes injection site reactions, influenza-like symptoms, infection, fever, tumor, cardiovascular event，drug-induced liver and kidney damage.

CONTACTS AND LOCATIONS:
Overall Officials: Sirui Yang, MD and PhD, Principal Investigator — The First Hospital of Jilin University
Locations (1):
- Sirui Yang, Changchun, Changchun/Jilin, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Rosenzwajg M, Lorenzon R, Cacoub P, Pham HP, Pitoiset F, El Soufi K, RIbet C, Bernard C, Aractingi S, Banneville B, Beaugerie L, Berenbaum F, Champey J, Chazouilleres O, Corpechot C, Fautrel B, Mekinian A, Regnier E, Saadoun D, Salem JE, Sellam J, Seksik P, Daguenel-Nguyen A, Doppler V, Mariau J, Vicaut E, Klatzmann D. Immunological and clinical effects of low-dose interleukin-2 across 11 autoimmune diseases in a single, open clinical trial. Ann Rheum Dis. 2019 Feb;78(2):209-217. doi: 10.1136/annrheumdis-2018-214229. Epub 2018 Nov 24. PMID 30472651
- [Background] Fontenot JD, Rasmussen JP, Gavin MA, Rudensky AY. A function for interleukin 2 in Foxp3-expressing regulatory T cells. Nat Immunol. 2005 Nov;6(11):1142-51. doi: 10.1038/ni1263. Epub 2005 Oct 16. PMID 16227984
- [Background] Malek TR. The biology of interleukin-2. Annu Rev Immunol. 2008;26:453-79. doi: 10.1146/annurev.immunol.26.021607.090357. PMID 18062768
- [Background] Cheng G, Yu A, Malek TR. T-cell tolerance and the multi-functional role of IL-2R signaling in T-regulatory cells. Immunol Rev. 2011 May;241(1):63-76. doi: 10.1111/j.1600-065X.2011.01004.x. PMID 21488890